CLINICAL TRIAL: NCT04952012
Title: The Effect of Thyroid Antibodies on Female Reproductive Function and Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First People's Hospital of Yuhang (Unknown); Taizhou Women and Children's Hospital Affiliated to Wenzhou Medical University (Unknown); Changxing People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-678
Record Dates: First submitted 2021-06-20; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-11

CONDITIONS: Thyroiditis, Autoimmune
MeSH Terms: conditions — Thyroiditis, Autoimmune

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ATA-positive
  Interventions: Drug: LT4
- ATA-negative
  Interventions: Drug: LT4

INTERVENTIONS:
Drug: LT4 — LT4 is used to improve the thyroid function of pregnant women.

SUMMARY:
Some women at reproductive age have positive antithyroid antibodies (ATAs). Thyroid peroxidase antibody (TPOAb) and thyroglobulin antibody (TgAb) are the most common ATAs. This study aimed to evaluate the impact of ATAs on maturation of women reproductive system and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age during 18-45y;
* Women tested for TPOAb and/or TgAb, TSH, free T3, free T4, total T3 and total T4 during the 1st trimester of pregnancy

Exclusion Criteria:

* Multiple pregnancies;
* Age < 18 y or > 40 y;
* L-T4 or PTU intervention before pregnancy;
* Other autoimmune diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects were all in the 1st trimester of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of pregnancy complications in women with or without thyroid antibodies | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China